CLINICAL TRIAL: NCT03974178
Title: Efficacy and Safety of Fexinidazole in Patients With Human African Trypanosomiasis (HAT) Due to Trypanosoma Brucei Rhodesiense: a Multicentre, Open-label Clinical Trial
Brief Title: Fexinidazole in Human African Trypanosomiasis Due to T. b. Rhodesiense
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-FEX-07-HAT
Record Dates: First submitted 2019-05-23; First posted 2019-06-04 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Trypanosomiasis, African; Sleeping Sickness; Trypanosoma Brucei Rhodesiense; Infection
Keywords: Trypanosoma Brucei (T. b.) rhodesiense; HAT; Neglected Tropical Disease
MeSH Terms: conditions — Trypanosomiasis, African; Infections; Neglected Diseases | interventions — fexinidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with stage 1 r-HAT (Experimental): Patients with stage 1 r-HAT were patients without trypanosomes in the cerebrospinal fluid (CSF) but with trypanosomes in the blood and/or lymph and CSF white blood cells (WBC) ≤5 cells/µL. Patients were to receive fexinidazole orally for 10 days.
  Interventions: Drug: Fexinidazole
- Patients with stage 2 r-HAT (Experimental): Patients with stage 2 r-HAT were patients with trypanosomes in the CSF (and/or in blood/lymph) and/or CSF WBC >5 cells/µL. Patients were to receive fexinidazole orally for 10 days.
  Interventions: Drug: Fexinidazole

INTERVENTIONS:
Drug: Fexinidazole — Tablets of 600 mg; Participants with a weight between 20 and 34 kg received 1200 mg (2 tablets) for 4 days, then 600 mg (1 tablet) for 6 days (with food); Participants with a weight of 35 kg and above received 1800 mg (3 tablets) for 4 days, then 1200 mg (2 tablets) for 6 days (with food)

SUMMARY:
The ultimate goal of this study is to show that fexinidazole offers an alternative over the existing treatments of Human African trypanosomiasis due to Trypanosoma brucei rhodesiense (r-HAT): melarsoprol in patients with stage 2 r-HAT and suramin in patients with stage 1 r-HAT. The main questions it aims to answer are:

* Is the short-term fatality rate and failure rate associated with fexinidazole lower than those of melarsoprol in patients with stage 2 r-HAT?
* Is the long-term failure rate associated with fexinidazole lower than that of melarsoprol in patients with stage 2 r-HAT?
* Can fexinidazole in patients with stage 1 r-HAT replace the treatment with suramin?
* Is fexinidazole treatment safe in patient with r-HAT, regardless of stage?

Participants will receive fexinidazole oral treatment for 10 days. Regular blood draws and lumbar punctures will be performed over 12 months to confirm the cure of the disease. Other assessments will include the recording of adverse events, signs and symptoms of the disease, laboratory tests, vital signs, electrocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (plus assent for children)
* ≥ 6 years old
* ≥ 20 kg body weight
* Ability to ingest at least one complete meal per day (or at least one Plumpy'Nut® sachet)
* Karnofsky index ≥ 40
* Parasitological confirmation of T. b. rhodesiense infection
* Having a permanent address or being traceable by others and willing and able to comply with follow-up visit schedule
* Agreement to be hospitalised for a minimum of 13 days and to receive the study treatment

Exclusion Criteria:

* Active clinically relevant medical conditions other than HAT that may jeopardize subject safety or at the investigator discretion may interfere with participation in the study.
* Compromised general health or severely deteriorated general condition, such as severe malnutrition, cardiovascular shock, respiratory distress, or terminal illness
* Patients with severe hepatic impairment (e.g.: clinical signs of cirrhosis or jaundice)
* Known hypersensitivity to fexinidazole, to any nitroimidazole drugs (e.g. metronidazole, tinidazole), or to any of the excipients
* Patients previously enrolled in the study or having already received fexinidazole

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enock Matovu, Prof, Principal Investigator — Makerere University
Locations (2):
- Rumphi District Hospital, Rumphi, Malawi
- Lwala Hospital, Lwala, Kadeberamaido, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matovu E, Nyirenda W, Eriatu A, Alves D, Perdrieu C, Lemerani M, Wamboga C, Lejon V, Seixas J, Signorell A, Reymondier A, Baudin E, Scherrer B, Valverde Mordt O. Fexinidazole as a new oral treatment for human African trypanosomiasis due to Trypanosoma brucei rhodesiense: a prospective, open-label, single-arm, phase 2-3, non-randomised study. Lancet Glob Health. 2025 May;13(5):e910-e919. doi: 10.1016/S2214-109X(25)00016-6. PMID 40288400

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 1 center in Malawi (Rumphi District Hospital) and 1 center in Uganda (Lwala Hospital). 46 participants were screened and signed informed consent. The screening pool was enlarged to other hospitals and centres in Uganda, Rumphi/Mzimba North District (Malawi), and Nkhotakota District (Malawi), from where patients could be referred to Lwala and Rumphi Hospitals for treatment. 45 participants were enrolled between 29 Sep 2019 and 17 Nov 2021.
Pre-assignment Details: The pre-treatment period of up to 7 days included screening and treatment of concurrent malaria and soil-transmitted helminthiasis. At the end of this period, all participants were treated with fexinidazole, regardless of the stage of human African trypanosomiasis due to Trypanosoma brucei rhodesiense (r-HAT) and treatment setting.
Groups:
- Patients With Stage 1 r-HAT: Patients without trypanosomes in the CSF but with trypanosomes in the blood and/or lymph and CSF WBC ≤5 cells/µL were classified as stage 1.
  Fexinidazole: Tablets of 600 mg; Participants with a weight between 20 and 34 kg received 1200 mg (2 tablets) for 4 days, then 600 mg (1 tablet) for 6 days (with food); Participants with a weight of 35 kg and above received 1800 mg (3 tablets) for 4 days, then 1200 mg (2 tablets) for 6 days (with food).
- Patients With Stage 2 r-HAT: Patients with trypanosomes in the CSF (and/or in blood/lymph) and/or CSF WBC >5 cells/µL were classified as stage 2.
  Fexinidazole: Tablets of 600 mg; Participants with a weight between 20 and 34 kg received 1200 mg (2 tablets) for 4 days, then 600 mg (1 tablet) for 6 days (with food); Participants with a weight of 35 kg and above received 1800 mg (3 tablets) for 4 days, then 1200 mg (2 tablets) for 6 days (with food).
Period: Overall Study
Arm/Group | Patients With Stage 1 r-HAT | Patients With Stage 2 r-HAT
Started | 10 | 35
Completed | 10 | 34
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients who took at least one dose of fexinidazole
Groups:
- Patients With Stage 1 r-HAT: Patients with stage 1 r-HAT were patients without trypanosomes in the cerebrospinal fluid (CSF) but with trypanosomes in the blood and/or lymph and CSF white blood cells (WBC) ≤5 cells/µL.
- Patients With Stage 2 r-HAT: Patients with stage 2 r-HAT were patients with trypanosomes in the CSF (and/or in blood/lymph) and/or CSF WBC >5 cells/µL.
- Total: Total of all reporting groups
Arm/Group | Patients With Stage 1 r-HAT | Patients With Stage 2 r-HAT | Total
Number analyzed (Participants) | 10 | 35 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (18.3) | 25.2 (15.2) | 27.0 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 13 | 14
  Male | 9 | 22 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Sub-Saharan African | 10 | 35 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 9 | 34 | 43
  Uganda | 1 | 1 | 2
r-HAT stage: Stage 1, Stage 2 [Count of Participants; unit: Participants] — Patients with stage 1 r-HAT (early stage, or haemolymphatic stage) were patients without trypanosomes in the cerebrospinal fluid (CSF) but with trypanosomes in the blood and/or lymph and CSF white blood cells (WBC) ≤5 cells/µL.
  Patients with stage 2 r-HAT (late stage, or meningoencephalitic stage) were patients with trypanosomes in the CSF (and/or in blood/lymph) and/or CSF WBC >5 cells/µL.
  Participants
    Stage 1 | 10 | 0 | 10
    Stage 2 | 0 | 35 | 35
White blood cells (WBC) in cerebrospinal fluid (CSF) [Mean (Standard Deviation); unit: cells/µL] | 1.7 (1.6) | 79.3 (103.2) | 62.1 (96.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Evaluable Patients With Stage 2 r-HAT Who Died by the End of Hospitalization, Considering Only Deaths Possibly Related to r-HAT or Fexinidazole
Description: The percentage of patients who died between the first intake of fexinidazole until the End-of-Hospitalization Visit (Day 12-18), considering only deaths possibly related to r-HAT or study treatment as assessed by the Data Safety Monitoring Board (DSMB), was calculated. The World Health Organization(WHO) verbal autopsy questionnaire was used since anatomopathological techniques were not available at the study sites (unless the death occurred at the hospital, in which case the investigator was present). In case of death that was not related to r-HAT nor to the study treatment during the hospitalization, the patient is considered as non-evaluable for efficacy purposes. Any patient who left the hospital without being medically discharged by the site Investigator before the planned End-of-Hospitalization Visit, and for whom no outcome could be retrieved, is also to be considered as non-evaluable.
Time Frame: 12 to 18 days after start of treatment
Population: The analysis is performed in evaluable patients with stage 2 r-HAT. A total of 35 patients with stage 2 r-HAT were enrolled and treated. One patient died during hospitalization, but the death was considered unrelated to r-HAT and/or the study treatment, as evaluated by the Investigator and the DSMB and accepted by the Sponsor. As per protocol, this patient was considered non-evaluable for efficacy purposes. There were 34 patients with stage 2 r-HAT who were evaluable.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Patients With Stage 2 r-HAT
Number analyzed (Participants) | 34
percentage of participants | 0 [0 to 8.43]
Statistical Analysis 1: Comparison: Patients With Stage 2 r-HAT; The proportion of deaths (pdeath) is compared to the threshold of 8.5%, with H0 being pdeath = 8.5% or more. The 90% confidence interval of the fatality rate is calculated with the Clopper-Pearson method; Test type: Other — The minimal sample size to get a possible rejection of H0 (pdeath = 8.5% or more) in favour of H1 (pdeath <8.5%) was 34 evaluable patients with stage 2 r-HAT. The hypothesis was tested with a one-sided exact test for proportions at the 0.05 significance level; p = 0.0488, one-sided exact test — The rate of deaths possibly related to r-HAT or to fexinidazole at the end of hospitalization was compared to the predefined unacceptable rate of 8.5%; Clopper Pearson exact method; Fatality rate = 0, 90% CI 2-sided [0 to 8.43]

2. Secondary Outcome: Percentage of Evaluable Patients With Stage 2 r-HAT, Whose Treatment Outcome is a Failure at the End of Hospitalization
Description: Treatment outcome at end of hospitalization (Day 12-18) is categorized as success or failure. Failure is defined as any of the following: presence of trypanosomes in any body fluid at end of treatment (Day 11), death related to r-HAT or fexinidazole at end of hospitalization according to the DSMB, or absence of clinical improvement leading to the use of rescue medication. Unrelated deaths are neither success nor failure (the patient is considered non-evaluable for efficacy purposes).
Time Frame: 12 to 18 days after start of treatment
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Patients With Stage 2 r-HAT
Number analyzed (Participants) | 34
percentage of participants | 0 [0 to 8.43]
Statistical Analysis 1: Comparison: Patients With Stage 2 r-HAT; The proportion of failures at the end of hospitalization (pfailure) is compared to the threshold of 9%, with H0 being pfailure = 9% or more. The 90% confidence interval of the failure rate is calculated with the Clopper-Pearson method; Test type: Other — The hypothesis H0 (pfailure at the end of hospitalization = 9% or more) was tested with a one-sided exact test for proportions at the 0.05 significance level; p = 0.0405, one-sided exact test — The rate of failures at the end of hospitalization was compared to the predefined unacceptable rate of 9%; Clopper Pearson exact method; Failure rate = 0, 90% CI 2-sided [0 to 8.43]

3. Secondary Outcome: Percentage of Evaluable Patients With Stage 2 r-HAT, Whose Treatment Outcome is a Failure at 12 Months
Description: Treatment outcome at test of cure (Month 12) is categorized as success or failure. Failure is defined as any of the following: presence of trypanosomes in any body fluid, death related to r-HAT or fexinidazole according to the DSMB, absence of clinical improvement leading to the use of rescue medication, or WBC count in the CSF >20 cells/μL which was unlikely due to causes other than HAT. Unrelated deaths are neither success nor failure (the patient is considered non-evaluable for efficacy purposes).
Time Frame: 12 months after start of treatment
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Patients With Stage 2 r-HAT
Number analyzed (Participants) | 34
percentage of participants | 2.94 [0.15 to 13.21]
Statistical Analysis 1: Comparison: Patients With Stage 2 r-HAT; The proportion of failures at 12 months (pfailure) is compared to the threshold of 12%, with H0 being pfailure = 12% or more. The 90% confidence interval of the failure rate is calculated with the Clopper-Pearson method; Test type: Other — The hypothesis H0 (pfailure at 12 months = 12% or more) was tested with a one-sided exact test for proportions at the 0.05 significance level; p = 0.0730, one-sided exact test — The rate of failures at 12 months was compared to the predefined unacceptable rate of 12%; Clopper Pearson exact method; Failure rate = 2.94, 90% CI 2-sided [0.15 to 13.21]

4. Secondary Outcome: Percentage of Evaluable Patients With Stage 1 r-HAT, Whose Treatment Outcome is a Failure at the End of Hospitalization
Description: as for outcome 2
Time Frame: 12 to 18 days after start of treatment
Population: The analysis is performed in evaluable patients with stage 1 r-HAT. None of patients with stage 1 r-HAT died from causes related to r-HAT or study treatment; therefore, all 10 patients were evaluable. Because the number of patients with stage 1 r-HAT is very small, no null hypotheses are testable and only descriptive data are provided.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Stage 1 r-HAT
Number analyzed (Participants) | 10
percentage of participants | 0

5. Secondary Outcome: Percentage of Evaluable Patients With Stage 1 r-HAT, Whose Treatment Outcome is a Failure at 12 Months
Description: as for outcome 3
Time Frame: 12 months after start of treatment
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Stage 1 r-HAT
Number analyzed (Participants) | 10
percentage of participants | 0

6. Secondary Outcome: Percentage of Evaluable Patients With Any r-HAT Stage Who Died by the End of Hospitalization, Considering Only Deaths Possibly Related to r-HAT or Fexinidazole
Description: The percentage of patients who died between the first intake of fexinidazole until the End-of-Hospitalization Visit (Day 12-18), considering only deaths possibly related to r-HAT or study treatment as assessed by the DSMB, was calculated. The WHO verbal autopsy questionnaire was used since anatomopathological techniques were not available at the study sites (unless the death occurred at the hospital, in which case the investigator was present). In case of death that was not related to r-HAT nor to the study treatment during the hospitalization, the patient is considered as non-evaluable for efficacy purposes. Any patient who left the hospital without being medically discharged by the site Investigator before the planned End-of-Hospitalization Visit, and for whom no outcome could be retrieved, is also to be considered as non-evaluable.
Time Frame: 12 to 18 days after start of treatment
Population: The analysis is performed in evaluable patients with any r-HAT stage. A total of 45 patients were enrolled and treated. One patient died during hospitalization, but the death was considered unrelated to r-HAT and/or the study treatment, as evaluated by the Investigator and the DSMB and accepted by the Sponsor. As per protocol, this patient was considered non-evaluable for efficacy purposes. There were 44 patients who were evaluable.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Patients With Any r-HAT Stage: Patients with any r-HAT stage, who were to receive fexinidazole orally for 10 days
Arm/Group | Patients With Any r-HAT Stage
Number analyzed (Participants) | 44
percentage of participants | 0 [0 to 6.58]
Statistical Analysis 1: Comparison: Patients With Any r-HAT Stage; [analysis description as in outcome 1, analysis 1]; Test type: Other — The hypothesis H0 (pdeath = 8.5% or more) was tested with a one-sided exact test for proportions at the 0.05 significance level; p = 0.0201, one-sided exact test — [p-value comment as in outcome 1, analysis 1]; Clopper Pearson exact method; Fatality rate = 0, 90% CI 2-sided [0 to 6.58]

7. Secondary Outcome: Percentage of Evaluable Patients With Any r-HAT Stage, Whose Treatment Outcome is a Failure at the End of Hospitalization
Description: as for outcome 2
Time Frame: 12 to 18 days after start of treatment
Population: as for outcome 6
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Patients With Any r-HAT Stage
Number analyzed (Participants) | 44
percentage of participants | 0 [0 to 6.58]
Statistical Analysis 1: Comparison: Patients With Any r-HAT Stage; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0158, one-sided exact test — The rate of failures at the end of hospitalization was compared to the predefined unacceptable rate of 9%; Clopper Pearson exact method; Failure rate = 0, 90% CI 2-sided [0 to 6.58]

8. Secondary Outcome: Percentage of Evaluable Patients With Any r-HAT Stage, Whose Treatment Outcome is a Failure at 12 Months
Description: as for outcome 3
Time Frame: 12 months after start of treatment
Population: as for outcome 6
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Patients With Any r-HAT Stage
Number analyzed (Participants) | 44
percentage of participants | 2.27 [0.12 to 10.34]
Statistical Analysis 1: Comparison: Patients With Any r-HAT Stage; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.0253, one-sided exact test — The rate of failures at 12 months was compared to the predefined unacceptable rate of 12%; Clopper Pearson exact method; Failure rate = 2.27, 90% CI 2-sided [0.12 to 10.34]

9. Secondary Outcome: Number of Participants With Any AE (Including Abnormal Laboratory or ECG Finding if Considered Clinically Significant) Until the End of Hospitalization
Description: Treatment-emergent AEs during the observation period were recorded from the first intake of fexinidazole (Day 1) until the End-of-Hospitalization Visit (between Day 12 and Day 18).
Time Frame: 12 to 18 days (between Day 1 and Day 12-18)
Population: The analysis is performed in all patients who took at least one dose of fexinidazole (regardless of r-HAT stage).
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Any r-HAT Stage
Number analyzed (Participants) | 45
Participants | 22

10. Secondary Outcome: Number of Participants With Any AE Considered as Serious Until the End of the Follow-up Period
Description: Treatment-emergent AEs considered as serious were collected from the first intake of fexinidazole (Day 1) until the End-of-Study Visit (Month 12). An AE was considered as serious if resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly or birth defect, or was an important medical event.
Time Frame: 12 months (between Day 1 and Month 12)
Population: The analysis is performed in all patients who took at least one dose of fexinidazole (regardless of r-HAT stage).
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Any r-HAT Stage
Number analyzed (Participants) | 45
Participants | 3

11. Secondary Outcome: Number of Participants With Any AE Considered as Possibly Related to Fexinidazole Until the End of the Follow-up Period
Description: Treatment-emergent AEs considered as possibly related to fexinidazole were collected from the first intake of fexinidazole (Day 1) until the End-of-Study Visit (Month 12).
Time Frame: 12 months (between Day 1 and Month 12)
Population: The analysis is performed in all patients who took at least one dose of fexinidazole (regardless of r-HAT stage).
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Any r-HAT Stage
Number analyzed (Participants) | 45
Participants | 5

ADVERSE EVENTS:
Time Frame: Non-serious treatment-emergent adverse events (AEs) were recorded from the first intake of fexinidazole (Day 1) until the End-of-Hospitalization Visit (Day 12-18). Treatment-emergent AEs considered as serious or related to fexinidazole treatment were collected from the first intake of fexinidazole (Day 1) until the End-of-Study Visit (Month 12). The population of analysis includes all patients who received at least one dose of fexinidazole.
Description: Adverse events were classified as serious according to the standard definition. In addition, in this study, alanine aminotransferase or aspartate aminotransferase levels higher than 3 times the upper limit of normal associated with total bilirubin levels higher than 2 times the upper limit of normal were considered as serious AEs (SAEs). Furthermore, any suspected transmission of an infectious agent via a medicinal product was also considered as an SAE.
Arm/Group | Patients With Stage 1 r-HAT | Patients With Stage 2 r-HAT
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/35
Serious Adverse Events (participants affected / at risk) | 0/10 | 3/35
Other Adverse Events (participants affected / at risk) | 6/10 | 16/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Stage 1 r-HAT (N=10) | Patients With Stage 2 r-HAT (N=35)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Stage 1 r-HAT (N=10) | Patients With Stage 2 r-HAT (N=35)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Electrocardiogram U-wave abnormality (Investigations) | 1 (1) | 2 (3)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Malaria (Infections and infestations) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The main limitation is the benchmark study design. A direct comparison with melarsoprol was impossible due to its toxicity (5% of patients die due to treatment-related encephalopathy) and the rarity of r-HAT cases. The annual number of r-HAT cases in all endemic countries decreased from 110 patients in 2012 to 27 in 2017. Although the primary endpoint required a subjective assessment of the cause of death, this was performed by independent experts from the safety committee to ensure robustness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor authorizes publications by a single site provided that multicentric results are published beforehand and that any communication is submitted to sponsor for review at least 28 days ahead of the expected date of publication. Upon sponsor request, any confidential information will have to be removed from the communication before publishing.

DOCUMENTS (2):
  • Study Protocol (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT03974178/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT03974178/SAP_001.pdf